CLINICAL TRIAL: NCT03276663
Title: Effect of a New Formula With a Reduced Concentration of Partially Hydrolyzed Protein on Growth of Healthy Term Infants: an Open-label Study
Brief Title: Growth of Healthy Term Infants Fed a Partially Hydrolyzed Follow-up Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15.01.INF
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Growth

STUDY DESIGN:
Intervention Model Description: Open-label, two-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formula fed group (Other): Formula feeding regimen
  Interventions: Other: Formula feeding regimen
- Human milk-fed group (No Intervention)

INTERVENTIONS:
Other: Formula feeding regimen — The feeding regimen consists of an existing commercial starter formula followed by a new follow-up formula
  Arms: Formula fed group

SUMMARY:
Growth of healthy term formula-fed infants who receive a single feeding regimen consisting of an existing partially hydrolyzed starter formula, then subsequently fed a partially hydrolyzed follow-up formula over the first year of life.

ELIGIBILITY:
Inclusion criteria:

1. Having obtained his/her parents' (or his/her legally accepted representative's [LAR's]) written informed consent and having evidence of personally signed and dated informed consent document indicating that the infant's parents/LAR have been informed of all pertinent aspects of the study.
2. Age ≤ 14 days after birth (date of birth = Day 0).
3. Full-term gestational birth (≥ 37 and ≤ 42 weeks).
4. Weight at birth ≥ 2500 g and ≤ 4200 g
5. Born to mothers with (normal) pre-pregnancy BMI ≥ 18.5 to < 26 kg/m2.
6. For formula-fed infants: born to mothers who independently elected, before study enrollment, not to breastfeed, but having received any HM is permitted (not applicable for infants in the HM-fed group)
7. For HM-fed infants: mothers intend to provide breast milk until age 6 months
8. Infant's parent(s)/LAR is of legal age of consent, has sufficient command of the French language to complete the informed consent and other study documents, and is willing and able to fulfill the requirements of the study protocol.
9. Infant's parent(s)/LAR is able to be contacted directly by telephone throughout the study.

Exclusion criteria:

1. Born to mothers with hormonal or metabolic disease (e.g. Type-1, Type-2, or gestational diabetes diagnosed according to standardized criteria).
2. Born to mothers who smoked > 10 cigarettes per day during pregnancy.
3. Born to mothers who used illicit drugs (e.g. marijuana, cocaine, amphetamines, or heroin) or alcohol (> 3 alcoholic beverages per week) during pregnancy.
4. Cognitive or physical developmental disorders (e.g., malabsorptive disorders such as short bowel syndrome; neurological and congenital disorders that may delay growth such as cerebral palsy, agenesis of the corpus callosum, spina bifida, Down syndrome, Cri Du Chat; disorders that may lead to obesity such as Prader Willi syndrome, Angelman syndrome; other renal, hepatic, pancreatic, or cardiovascular disorders).
5. Participation in any other clinical trial prior to enrollment.
6. Infants or infant's family who in the Investigator's judgment cannot be expected to comply with the protocol or study procedures.

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 194 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Growth velocity (weight gain in g/day) of healthy term formula-fed infants during the first 6 months | 6 month
  compared to the WHO reference standards or to the human milk (HM)-fed comparator group.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Billeaud, Principal Investigator — University Hospital, Bordeaux
Locations (6):
- France (6):
  - CHU Amiens Picardie Site SUD, Amiens
  - CHU Bordeaux - Hôpital Pellegrin Enfants, Bordeaux
  - CHU de Caen, Caen
  - CHU Nantes - Hôpital Mère-Enfant, Nantes
  - Hopital Necker, Paris
  - Biofortis CIC, Saint-Herblain

REFERENCES:
- [Derived] Billeaud C, Adamon L, Piloquet H, Hays NP, Dupuis L, Metreau I, Leke A. A new partially hydrolyzed whey-based follow-on formula with age-adapted protein content supports healthy growth during the first year of life. Front Pediatr. 2022 Sep 28;10:937882. doi: 10.3389/fped.2022.937882. eCollection 2022. PMID 36245743